CLINICAL TRIAL: NCT06840470
Title: Investigating the Effect of Topical Imiquimod on Sebaceous Hyperplasia
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Sunny Wong, Associate Professor of Dermatology, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM00262234
Record Dates: First submitted 2025-02-17; First posted 2025-02-21 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Sebaceous Hyperplasia
Keywords: Lesions on both sides of the face; Topical imiquimod
MeSH Terms: interventions — Imiquimod

STUDY DESIGN:
Intervention Model Description: Each subject's face will be divided randomly into an imiquimod-treated side and an untreated control side.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Imiquimod (Experimental): Will be applied 3 times weekly ((i.e. Monday, Wednesday, and Friday prior to bedtime) to one side of the face.
  Interventions: Drug: Imiquimod 5% Topical Cream
- No treatment (No Intervention): Lesions on the other side of the face will not be treated. Participants will have baseline and follow-up visits that will include photographs of the lesions.

INTERVENTIONS:
Drug: Imiquimod 5% Topical Cream — Participants will apply this cream to one side of the face 3 times a week for up to 8 weeks. The cream will be applied before bedtime. The imiquimod should be washed off with mild soap and water after 6-10 hours. Participants will have baseline and follow-up visits that will include photographs of the lesions.
  Other Names: Aldara
  Arms: Imiquimod

SUMMARY:
This study is being completed to determine if 8 weeks of treatment with imiquimod can shrink sebaceous hyperplasia.

ELIGIBILITY:
Inclusion Criteria:

* Patient has sebaceous hyperplasia lesions on both sides of the face. At least one sebaceous hyperplasia lesion on each side of the face is 1 mm or more in size.
* If of child-bearing potential, subject agrees to the use of highly effective contraception during study participation. For women of childbearing potential, acceptable pregnancy prevention measures will include abstinence, barrier methods, chemical methods, or surgical.
* Ability to understand and willingness to sign a written informed consent

Exclusion Criteria:

* Current use or prior use of a retinoid (e.g. tretinoin) within the last 4 weeks.
* Prior use of imiquimod on the treated area.
* Concurrent use of 5-fluorouracil, aminolevulinic acid (photodynamic therapy), or psoralen therapy, or use of any of these within the last 4 weeks.
* Concurrent facial peels or cosmetic laser therapy on the treated areas.
* Nursing, pregnant or planning to become pregnant.
* Immunocompromised status (e.g. organ transplantation recipients or patients on cyclosporine).
* Current participation in other investigational trials.
* Known or suspected history of a clinically significant systemic disease (e.g., immunological deficiencies), unstable medical disorders (e.g., unstable diabetes), life-threatening disease or current malignancies.
* Known hypersensitivity to any of the following (in any dosage form): imiquimod or any component of the study medications.
* Received radiation therapy and/or anti-neoplastic agents within 3 months prior to study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-03-11 (Actual); Primary Completion 2027-03-11 (Estimated); Study Completion 2027-09-11 (Estimated)

PRIMARY OUTCOMES:
Complete and 75% clearance rates (clearance refers to reduction in total lesional area) at 16 weeks of treated lesions | 16 weeks

SECONDARY OUTCOMES:
Mean change in Sebaceous Hyperplasia (SH) count | 16 weeks
Mean change in Sebaceous Hyperplasia (SH) diameter | 16 weeks
Adverse events (AE) associated with imiquimod 5% cream when used in the treatment of sebaceous hyperplasia | Up to 8 weeks
  The following will be described for Adverse events per protocol:
  * Serious or non-serious
  * Mild, moderate, Severe
  * The relationship (unexpected or expected) of the study drug
  * Attribution of the AE: Definite, Probably, Possible, Unlikely, Unrelated.

CONTACTS AND LOCATIONS:
Overall Officials: Sunny Wong, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No